CLINICAL TRIAL: NCT05104970
Title: Comparative Pharmacokinetics of Two Different Oral Delivery Systems of Cholecalciferol
Acronym: PLUTO
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Scotmann Pharmaceuticals (Industry)
Collaborators: Rawalpindi Medical College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SunnyD
Record Dates: First submitted 2021-10-26; First posted 2021-11-03 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Vitamin D Deficiency
Keywords: Vitamin D
MeSH Terms: conditions — Vitamin D Deficiency

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: double blinded placebo controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- SunnyD STAT softgel capsule (Active Comparator): Cholecalciferol 200000 IU
  Interventions: Dietary Supplement: SunnyD STAT softgel capsule
- Placebo SunnyD STAT softgel capsule (Placebo Comparator): Olive oil only
  Interventions: Dietary Supplement: Placebo SunnyD STAT softgel capsule
- SunnyD insta ampoule (Active Comparator): Vitamin D3 200000 IU
  Interventions: Drug: SunnyD insta ampoule
- Placebo SunnyD insta ampoule (Placebo Comparator): Olive oil only
  Interventions: Drug: Placebo SunnyD insta ampoule

INTERVENTIONS:
Drug: SunnyD insta ampoule — Cholecalciferol 200000 IU insta ampoule
  Arms: SunnyD insta ampoule
Dietary Supplement: SunnyD STAT softgel capsule — Cholecalciferol 200000 IU softgel capsule
  Arms: SunnyD STAT softgel capsule
Drug: Placebo SunnyD insta ampoule — Olive oil
  Arms: Placebo SunnyD insta ampoule
Dietary Supplement: Placebo SunnyD STAT softgel capsule — Olive oil
  Arms: Placebo SunnyD STAT softgel capsule

SUMMARY:
The aim of this study is to adapt the gold standard of research and to explore the comparative bioavailability and clinical efficacy of the two most commonly used forms of Cholecalciferol i.e. ampoules and softgel capsules.

DETAILED DESCRIPTION:
Deficiency of Vitamin D is highly prevalent in all sectors and regions of Pakistan. Its effects encompass multiple pluripotent physiological impacts on human body, including its classical action on bone health and immune modulation. Health care workers are routinely prescribing supplementations to correct the deficiencies. Different forms of Cholecalciferol are available in the market. It ranges from absorba liquids, drops, tablets, softgels to injectable and oral ampoules. Different delivery systems offer different advantages, challenges and efficacies specific to their specific pharmacokinetics. The aim of this study is to adapt the gold standard of research and to explore the comparative bioavailability and clinical efficacy of the two most commonly used forms of Cholecalciferol i.e. ampoules and softgel capsules.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Adult (20-70 years of age)
2. Vitamin D deficiency (serum 25(OH)D < 20 ng/ml)
3. Permanent employees of Medicine ward of Holy Family Hospital, DHQ, BBH hospitals and RMU for easy follow up throughout the study duration
4. Willingness and availability to show-up in the follow up visit and serum testing throughout the study period as needed

EXCLUSION CRITERIA:

1. Vitamin D sufficiency or moderate deficiency (serum 25(OH)D > 20 ng/ml)
2. Pregnant ladies
3. Participants already taking Vitamin D supplementation, anti-convulsants, barbiturates or steroids
4. Subjects with granulomatous conditions, liver disease, kidney disease, or diabetes

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-08-09 (Estimated); Primary Completion 2023-01-09 (Estimated); Study Completion 2023-02-10 (Estimated)

PRIMARY OUTCOMES:
Area Under Curve (AUC) | 70 days
  Area Under Curve (AUC) trail follow-up at 0,1,7,28,70. Trapezoidal method for calculations would be used and levels would be reported from lab essay of 25(OH)D

SECONDARY OUTCOMES:
Serum 25(OH)D level | 3 months
  Serum 25(OH)D level would be checked at the end of the trial after 3 months to assess the change in levels (if any). It would be assessed through laboratory essay

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Umar, MBBS,FCPS, Principal Investigator — Rawalpindi Medical College

IPD SHARING:
Plan to Share IPD: No
Proforma